CLINICAL TRIAL: NCT04618237
Title: Observational Study of Long-Term Joint Health Outcome in Hemophilia Patient
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Taipei Medical University Hospital (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: N202001021
Record Dates: First submitted 2020-09-23; First posted 2020-11-05 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-09

CONDITIONS: Hemophilia; Arthropathy
MeSH Terms: conditions — Hemophilia A; Joint Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Sample will be kept in ultra low temp. freezer and given subject numbers as identifiers.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients with severe hemophilia A can experience repeated bleeding into the same joint (ie, a target joint; most frequently in the ankle, knee, and elbow), which can contribute to hemophilic arthropathy and, over time, ultimately result in chronic pain, functional limitations, deformities, reduced joint of motion and decreased quality of life.

Early use of prophylaxis is recommended following diagnosis of severe hemophilia A to maintain joint health and prevent joint destruction. Eloctate is produced using a human cell line and an addition of an Fc fusion protein to recombinant FVIII (rFVIIIFc) with prolonged half-life and was launched in Taiwan from Nov. 2018. The pivotal studies of rFVIIIFc show that patients maintained a low bleeding rate, with most experiencing a median annualized bleeding rate (ABR) of 0 and 97% of target joints were resolved across adult, adolescent, and pediatric subjects during 4 years of prophylaxis rFVIIIFc treatment. However, in Taiwan we are still lacking the real world treatment outcome data on rFVIIIFc, especially for the joint health evidence in Asian Hemophilia A patients.

Therefore the objective of this study is to evaluate the effectiveness of rFVIIIFc treatment on joint health over a long observational period of 36 month focused on physical and functional changes in hemophilia A patients.

DETAILED DESCRIPTION:
Thermographic assessment has been proposed to be a potential tool in evaluating the inflammatory arthritis patients. Thermography has advantages of simple, time-saving, low skill demanding, no radiation exposure and non-invasiveness. It is possible to conduct a quantitative analysis with thermography. However, it is still unknown whether thermography evaluation can provide clinical information regarding the joint health in hemophilia arthropathy patients. The project will focus on:

1. Investigate the association among thermography findings and functional status in hemophilia arthroplasty
2. Investigate the novel biomarkers in predicting function in hemophilia arthropathy including: soft tissue ultrasound, body composition, thermographic findings of joints, muscle composition and serum biomarkers of joint degeneration.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to sign inform consent form and complied with study procedure
2. Patient received confirmative diagnosis of Hemophilia A Disease
3. Severe hemophilia A patient currently who are on treatment with Eloctate prior to enrolment visit (Note: Prescription based on physician's clinical judgement and discussion with patients)

Exclusion Criteria:

1. Unwilling to sign inform consent form.
2. History of major neurological disease (eg. Stroke, Parkinson's disease, neuropathy, etc.)
3. History of major psychiatric disease (eg. Schizophrenia, bipolar disorder)
4. Significantly impaired vision / hearing
5. Cannot communicate in Mandarin Chinese
6. Recent joint bleeding and trauma 3 months prior to study

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 35 severe Hemophilia A patients
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2020-07-20 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Hemophilia Joint Health Score (HJHS) | Baseline to 24 months follow up
  The HJHS measures joint health, in the domain of body structure and function (i.e. impairment), of the joints most commonly affected by bleeding in hemophilia: the knees, ankles, and elbows. The HJHS provides a total score (higher score is worse; max=124), joint specific scores, and a global gait score.
Musculoskeletal ultrasound/HEAD-US scoring system (Haemophilia Early Arthropathy Detection by UltraSound) | Baseline to 24 months follow up
  Musculoskeletal ultrasound could detect soft tissue alterations and be used as early detection of hemophilic arthropathy. Ultrasound assessment of bilateral knees and ankles, and bilateral gastrocnemius and quadriceps would be taken out in this study and scored with HEAD-US(Haemophilia Early Arthropathy Detection by UltraSound) scoring system. The scoring was based on three markers: synovitis (score 0-2), cartilage (score 0-4) and subchondral bone (score of 0-2) with a maximum score of eight points per joint, higher score is worse.
X-rays/Pettersson score (PS) | Baseline to 24 months follow up
  X-rays are used to evaluate structural changes in joints of patients with hemophilic arthropathy. X-rays images of bilateral knees and ankles will be taken in this study and scored with Pettersson scoring system. The maximum possible score for a given joint is 13 points and higher score is worse.
Thermography | Baseline to 24 months follow up
  Infrared thermography could be a simple tool to detect early inflammation of joints and joint associated structures. FLIR ONE imaging camera is used to take thermal images.

SECONDARY OUTCOMES:
Hemophilia activities list (HAL) | Baseline to 24 months follow up
  The HAL measures the impact of hemophilia on self-perceived functional abilities in 7 domains, including Lying/sitting/kneeling/standing, Functions of the legs , Functions of the arms, Use of transportation, Self-care, Household tasks, Leisure activities and sports.
Hemophilia Quality of Life Questionnaire for Adults (HAEM-A-QOL) | Baseline to 24 months follow up
  The HAEM-A-QOL assess health-related quality of life in haemophilia patients with 10 domains, including physical health, feelings, view, sport& leisure, work& school, dealing, treatment, future, family planning, and partnership.
Quality of life assessment (EQ-5D) - Descriptive System | Baseline to 24 months follow up
  The EQ-5D measures generic health status with 2 components: descriptive system and visual analogue scale. The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression.
Quality of life assessment (EQ-5D) - Visual Analogue Scale (VAS) | Baseline to 24 months follow up
  The EQ-5D measures generic health status with 2 components: descriptive system and visual analogue scale. The visual analogue scale (VAS) records the patient's self-rated health on a vertical visual analogue scale
Serum markers: cartilage oligomeric matrix protein (COMP) | Baseline to 24 months follow up
  COMP is considered a marker of cartilage breakdown, and is diagnostic of arthritis and to correlate with the disease severity. Serum COMP level is indicative of the amount of joint damage in patients with hemophilic arthropathy.
Serum markers: chondroitin-sulphate aggrecan turnover 846 epitope (CS846) | Baseline to 24 months follow up
  CS846 is a sensitive biomarker reflecting degradation of cartilage and synovial tissues. Serum CS-846 levels is indicative of the amount of joint damage in patients with hemophilic arthropathy.
6 mins walk test | Baseline to 24 months follow up
  The 6 mins walk test (MWT) measures the distance an individual could walk over six minutes on a hard, flat surface. The test could be used as a performance-based measure of functional exercise capacity.
  Gait Analysis (RehaWatch): RehaWatch is based on inertial sensors that allow the quantitative measurement of the kinemetic variables

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No